CLINICAL TRIAL: NCT00628953
Title: A Randomized, Double-Blind, Parallel Group Multicenter Efficacy and Safety Phase IIB Pilot Study of Esomeprazole 40mg Bid Versus Placebo Bid in Adult Asthmatics Treated for 4 Months
Brief Title: Adult Asthmatics and Acid Reflux
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Tore Lind, MD - Nexium Medical Science Director, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SD-NEE-0003; D9611C00003
Record Dates: First submitted 2008-02-26; First posted 2008-03-05 (Estimated); Last update posted 2009-03-13 (Estimated); Status verified 2009-03

CONDITIONS: Asthma
Keywords: Asthma; Acid Reflux; Nexium; Esomeprazole
MeSH Terms: conditions — Asthma; Gastroesophageal Reflux | interventions — Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Esomeprazole
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Esomeprazole — 40mg twice a day
  Other Names: Nexium
  Arms: 1
Drug: Placebo — 40mg twice a day
  Arms: 2

SUMMARY:
The purpose of this study is to assess the efficacy and safety of Nexium in the treatment of subjects with persistent asthma believed to have acid reflux as a contributory factor to control of their asthma.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of asthma
* Forced Expiratory Volume and Peak Expiratory Flow as defined by the protocol
* Daily use of inhaled GCS and/or leukotriene pathway modifier for greater than 3 months.
* Severe heartburn 3 days/week during the run-in period.

Exclusion Criteria:

* Subjects with a history of 3 sinus infections treated with antibiotics in the year prior to Visit 1.
* Any other significant disease or pathology judged to be clinically significant by the investigator

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2002-10; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Effect on asthma symptoms as measured by changes in Peak Expiratory Flow morning & evening, Forced Expiratory Volume and asthma symptom scores | 4 weekly

SECONDARY OUTCOMES:
Safety as assessed by adverse event recording and clinical and laboratory measurements. | 4 weekly

CONTACTS AND LOCATIONS:
Overall Officials: Paula Fernstrom, Study Director — Nexium Global Product Director, AstraZeneca